CLINICAL TRIAL: NCT02720198
Title: A Randomized Trial Comparing Efficacy and Tolerability of Levomilnacipran Switch Versus Adjunctive Quetiapine in Major Depressive Disorder (MDD) With Inadequate Response to SSRIs
Brief Title: Levomilnacipran ER vs. Adjunctive Quetiapine for Adults With Inadequate Relief With SSRIs in MDD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Forest Laboratories (Industry); Institute for Advanced Medical Research, Alpharetta, GA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00064983
Record Dates: First submitted 2016-03-16; First posted 2016-03-25 (Estimated); Results first posted 2019-07-02 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Levomilnacipran; Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Levomilnacipran (Active Comparator): Levomilnacipran ER is switched from SSRI.
  Interventions: Drug: Levomilnacipran
- Quetiapine (Active Comparator): Quetiapine XR is added in addition to current SSRI.
  Interventions: Drug: Quetiapine

INTERVENTIONS:
Drug: Levomilnacipran — treating major depression. A flexible dose regime of levomilnacipran ER 20-120 mg/d mg per day starting at 20 mg/d on Days 1-2, increasing to 40 mg/d on Days 3-7 in week 1, then flexibly dosed between 40 mg/d -120 mg/d during weeks 2 through 8
  Other Names: Fetzima
  Arms: Levomilnacipran
Drug: Quetiapine — Quetiapine will be started at 50 mg/d on Day 1-2, increasing to 150 mg/d on Days 3-7 in Week 1 and then flexibly dosed between 150-300 mg/d during Weeks 1 through 8 along with their current antidepressant.
  Other Names: Seroquel
  Arms: Quetiapine

SUMMARY:
This study's primary objective is to compare the efficacy and tolerability of switching patients with inadequate relief on generic SSRIs to levomilnacipran versus adding a new treatment (quetiapine) to the participants' existing treatment with people diagnosed with depression (major depression disorder).

The secondary objective is to examine the response and remission rates following the switch from a generic SSRI to levomilnacipran ER and augmentation with quetiapine along with examining changes in neurocognitive and apathy measures after the switch.

DETAILED DESCRIPTION:
1. Study Design 1) An 8-week, randomized rater blinded parallel group, 2-arm trial 2) Trial duration - 9 weeks 3) Drug doses

   * Levomilnacipran ER; Switching to a flexible dose regime of levomilnacipran ER 40-120 mg/day after initial dose of 20mg.
   * Quetiapine XR; Adjunct a flexible dose regimen of quetiapine XR 150-300 mg/day after initial dose of 50mg.
2. Objective 1) To compare the efficacy and tolerability of switching to levomilnacipran ER (40-120 mg/d) versus augmentation with quetiapine XR 150-300 mg/day to the patients' existing treatment for patients with inadequate relief on generic SSRIs in patients with MDD.

2) To examine the response following the switch from generic SSRI to levomilnacipran ER and augmentation with quetiapine XR.

3) To examine changes in neurocognitive and apathy measures after switching from SSRI to levomilnacipran ER and after augmentation with quetiapine XR in MDD

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years inclusive
* Current diagnosis of MDD based on DSM-IV criteria
* Able to understand study rules and procedures and willing to sign written informed consent for study participation
* Inadequate response to antidepressants: having a score of ≥14 on the 17-item Hamilton Anxiety Scale (HAMD) and not having a ≥ 50% reduction in HAMD or CGI-S scores from baseline after a retrospective confirmation of an adequate trial of a single antidepressant (defined as a minimum 6-week trial of acceptable therapeutic dose (daily dose ≥ 40 mg of fluoxetine, 40 mg of paroxetine, 20 mg of citalopram, 10 mg of escitalopram, 37.5 mg of paroxetine CR, 150 mg of sertraline, 100 mg of fluvoxamine).
* If female, nonpregnant/nonlactating status
* Duration of current MDD ≥ 4 weeks and < 24 months
* Not more than 2 treatment failures of adequate antidepressant trials for current episode of MDD

Exclusion Criteria:

* Has previously participated in a levomilnacipran ER or quetiapine XR or quetiapine clinical study in previous 12 months

Has 1 or more the following:

* Current or past history of: manic or hypomanic episode, schizophrenia or any other psychotic disorder defined in the DSM- 5
* Diagnosis of alcohol or other substance use disorder (except nicotine and caffeine) as defined in the DSM-5 that has not been in sustained full remission for at least 6 months prior to screening (participant must also have negative urine drug screen prior to baseline).
* Presence or history of a clinically significant neurological disorder (including epilepsy)
* Poorly controlled Hypertension or Diabetes
* uncontrolled narrow-angle glaucoma
* hypersensitivity to levomilnacipran, milnacipran , quetiapine or quetiapine XR
* Neurodegenerative disorder.
* Has a thyroid stimulating hormone value outside the normal range at the Screening Visit that is deemed clinically significant by the investigator.
* Has clinically significant abnormal vital signs as determined by the investigator.
* Has a clinical significant abnormal electrocardiogram.
* Has screening laboratory values greater than 2.5 times the upper or lower limits of normal range or judged to be clinically significant
* Has a disease or takes medication that, in the opinion of the investigator, could interfere with the assessments of safety, tolerability, or efficacy or prevent the individual from completing the study.
* Female subjects of childbearing potential not on adequate contraception methods in the opinion of the investigator

  o If the female is childbearing, she must agree to use appropriate contraceptive measures for the duration of the study and for one month afterwards. Medically acceptable contraceptives include: (1) surgical sterilization (such as tubal ligation of hysterectomy), (2) approved hormonal contraceptives (such as birth control pills, patches, implants, or injections), (3) barrier methods (such as condom or diaphragm) used with a spermicide, or (4) an intrauterine device (IUD). Contraceptive measures such as Plan B ™, sold for emergency use after unprotected sex, are not acceptable methods for routine use. If the female does become pregnant during this study she must inform the study physician immediately.
* Has a significant risk of suicide according to Columbia Suicide Severity Rating Scale (CSSRS) or in the clinical judgment of the investigator
* History of suicide attempt in the previous 12 months
* MDD with postpartum onset, psychotic features or seasonal features
* Hamilton Anxiety Scale (HAM-A) baseline score ≥ 24
* Failure of ≥ 3 adequate trials of different antidepressants for the current episode of MDD
* ≥ 3 episodes major depression in previous 12 months or ≥ 8 lifetime episodes of MDD
* Current or previous use of an atypical or typical antipsychotic agent for augmentation of major depression or treatment of psychotic depression, mania psychosis, or agitation. Previous use of antipsychotics for insomnia will be permitted.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2018-06-12 (Actual); Study Completion 2018-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashwin A Patkar, MD, Principal Investigator — Duke Universtiy Medical Center
Locations (1):
- Institute for Advanced Medical Research, Alpharetta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential participants were identified by self-referral via the printed ad, phone script, the patients' physicians, local health providers, mental health providers, or Duke providers. Others were recommended by PI or Study Coordinator. They assessed and screened at 2 sites, an university hospital and a clinic of the research institute.
Pre-assignment Details: One subject was lost to follow up after screening.
Groups:
- Levomilnacipran: Levomilnacipran ER is switched from SSRI. Levomilnacipran ER: A flexible dose regime of levomilnacipran ER 20-120 mg/d mg per day, starting at 20 mg/d on Days 1-2, increasing to 40 mg/d on Days 3-7 in week 1, then flexibly dosed between 40 mg/d -120 mg/d during weeks 2 through 8.
- Quetiapine: Quetiapine XR was added in addition to current SSRI. Quetiapine XR: Quetiapine XR was started at 50 mg/d on Day 1-2, increasing to 150 mg/d on Days 3-7 in Week 1 and then flexibly dosed between 150-300 mg/d during Weeks 1 through 8 along with their current SSRI.
Period: Overall Study
Arm/Group | Levomilnacipran | Quetiapine
Started | 29 | 31
Completed | 29 | 30
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Levomilnacipran | Quetiapine | Total
Number analyzed (Participants) | 29 | 31 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 30 | 58
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.34 (14.28) | 46.13 (11.17) | 45.75 (12.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 9 | 11 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 29 | 30 | 59
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 25 | 45
  White | 9 | 4 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 29 | 31 | 60
Baseline SSRI [Count of Participants; unit: Participants]
  Escitalopram | 9 | 3 | 12
  Fluoxetine | 3 | 10 | 13
  Sertraline | 5 | 6 | 11
  Citalopram | 8 | 5 | 13
  Paroxetine | 3 | 7 | 10
  Unknown | 1 | 0 | 1
Baseline Dose of SSRI [Mean (Standard Deviation); unit: dose of medication, mg]
  mg(Escitalopram) | 18.89 (3.333) | 16.67 (5.774) | 18.33 (3.892)
  mg(Fluoxetine) | 53.33 (23.094) | 42.00 (6.325) | 44.62 (11.983)
  mg(Sertraline) | 170.00 (27.386) | 150.00 (31.623) | 159.09 (30.151)
  mg(Citalopram) | 21.25 (8.345) | 28.00 (10.954) | 23.85 (9.608)
  mg(Paroxetine) | 40.00 (0.000) | 51.43 (15.736) | 48.00 (13.984)

OUTCOME MEASURES:

1. Primary Outcome: Changes of Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score
Description: A ten-item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. Total scores will range from 0 to 60. Higher scores indicate greater severity of depressive episodes.
Time Frame: Baseline to Week 8
Population: Data not available on some participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Levomilnacipran | Quetiapine
Number analyzed (Participants) | 26 | 30
score on a scale | -5.81 (6.080) | -6.97 (7.632)
Statistical Analysis 1: Comparison: Levomilnacipran vs Quetiapine; Test type: Superiority; p = 0.53, t-test, 2 sided; Mean Difference (Final Values) = 1.159, 95% CI 2-sided [-2.518 to 4.836], Standard Error of Mean 1.834

2. Secondary Outcome: Response Rate
Description: Remission was defined as [>or=50% reduction in MADRS score with MADRS <or=10] and response was defined as [>or=50% reduction in MADRS with MADRS >10]. Response rate included remission and response.
Time Frame: Week 8
Population: Data not available on some participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Levomilnacipran | Quetiapine
Number analyzed (Participants) | 26 | 30
Participants | 3 | 7
Statistical Analysis 1: Comparison: Levomilnacipran vs Quetiapine; Test type: Superiority; p = 0.428, Mantel Haenszel; Odds Ratio (OR) = 0.492, 95% CI 2-sided [0.101 to 2.388], Standard Error of Mean 0.806

3. Secondary Outcome: Remission Rate
Description: Remission was defined as [>or=50% reduction in MADRS score with MADRS <or=10]
Time Frame: Week 8
Population: Data not available on some participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Levomilnacipran | Quetiapine
Number analyzed (Participants) | 26 | 30
Participants | 2 | 3
Statistical Analysis 1: Comparison: Levomilnacipran vs Quetiapine; Test type: Superiority; p = 0.272, Mantel Haenszel; Odds Ratio (OR) = 0.451, 95% CI 2-sided [0.109 to 1.866], Standard Error of Mean 0.724

4. Secondary Outcome: Changes in Neurocognition by Changes in Scores on Reyes Verbal Learning Test
Description: Number of words correctly recalled by the respondent is recorded. 1 point for each word correctly recalled. Total score range of 0-40. Higher scores mean better cognitive function.
Time Frame: Baseline to Week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Levomilnacipran | Quetiapine
Number analyzed (Participants) | 29 | 30
score on a scale | 2.28 (5.694) | 2.90 (5.255)
Statistical Analysis 1: Comparison: Levomilnacipran vs Quetiapine; Test type: Superiority; p = 0.664, t-test, 2 sided; Mean Difference (Final Values) = -0.624, 95% CI 2-sided [-3.484 to 2.236], Standard Error of Mean 1.428

5. Secondary Outcome: Changes in Neurocognition by Changes in Scores on Scores on Digit Symbol Substitution Test (DSST)
Description: DSST measures working memory and visuospatial processing. 1 point for each object correctly substituted from number to each matched symbol. Total score range of 0-89. Higher scores mean better cognitive function.
Time Frame: Baseline to Week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Levomilnacipran | Quetiapine
Number analyzed (Participants) | 29 | 30
score on a scale | 3.21 (9.321) | 0.87 (7.431)
Statistical Analysis 1: Comparison: Levomilnacipran vs Quetiapine; Test type: Superiority; p = 0.292, t-test, 2 sided; Mean Difference (Final Values) = 2.34, 95% CI 2-sided [-2.070 to 6.750], Standard Error of Mean 2.199

6. Secondary Outcome: Number of Subjects With Global Improvement in Scores on Clinical Global Impression Scale- Severity (CGI-S)
Description: CGI-S is a 7 point scale that assess the severity of illness and requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. It is used to assess the clinician's view of the patient's global functioning. Total score range of 0-7.
Time Frame: Baseline to Week 8
Measure: Count of Participants; unit: Participants
Arm/Group | Levomilnacipran | Quetiapine
Number analyzed (Participants) | 29 | 30
Participants | 13 | 13
Statistical Analysis 1: Comparison: Levomilnacipran vs Quetiapine; Test type: Superiority; p = 0.884, Mantel Haenszel; Odds Ratio (OR) = 1.063, 95% CI 2-sided [0.380 to 2.971], Standard Error of Mean 0.525

7. Secondary Outcome: Number of Subjects With General Improvement in Scores on Clinical Global Impression Scale- Improvement (CGI-I)
Description: CGI-I a 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. It is used to assess the clinician's view of the patient's global functioning. Total score range of 0-7.
Time Frame: Baseline to Week 8
Population: Data not available for some participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Levomilnacipran | Quetiapine
Number analyzed (Participants) | 27 | 30
Participants | 21 | 24
Statistical Analysis 1: Comparison: Levomilnacipran vs Quetiapine; Test type: Superiority; p = 0.905, Mantel Haenszel; Odds Ratio (OR) = 0.875, 95% CI 2-sided [0.245 to 3.129], Standard Error of Mean 0.650

8. Secondary Outcome: Changes of Anxiety Symptoms in Scores on Hamilton Anxiety Rating Scale (HAM-A)
Description: A questionnaire used by clinicians to rate the severity of a patient's anxiety. Total score range of 0-48. A higher score indicates greater anxiety.
Time Frame: Baseline to Week 8
Population: Data not available for all subjects.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Levomilnacipran | Quetiapine
Number analyzed (Participants) | 28 | 30
score on a scale | -3.89 (4.969) | -5.53 (5.859)
Statistical Analysis 1: Comparison: Levomilnacipran vs Quetiapine; Test type: Superiority; p = 0.254, t-test, 2 sided; Mean Difference (Final Values) = 1.64, 95% CI 2-sided [-1.211 to 4.492], Standard Error of Mean 1.423

9. Secondary Outcome: Changes of Quality of Life in Scores on Sheehan Disability Scale (SDS) Total
Description: A self-reported brief scale to assess impairment of work/school, social life and family and home. Total score range of 0-30. A higher score indicates greater impairment.
Time Frame: Baseline to Week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Levomilnacipran | Quetiapine
Number analyzed (Participants) | 29 | 30
score on a scale | -3.79 (6.477) | -0.10 (8.126)
Statistical Analysis 1: Comparison: Levomilnacipran vs Quetiapine; Test type: Superiority; p = 0.058, t-test, 2 sided; Mean Difference (Final Values) = -3.693, 95% CI 2-sided [-7.520 to 0.134], Standard Error of Mean 1.910

10. Secondary Outcome: Changes in Scores on Apathy Evaluation Scale (AES).
Description: Self-Administered assessment measuring lack of motivation not attributable to diminished level of consciousness, cognitive impairment, or emotional distress. Total scores range from 0-54. Higher scores indicate greater apathy.
Time Frame: Baseline to Week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Levomilnacipran | Quetiapine
Number analyzed (Participants) | 29 | 30
score on a scale | -2.07 (8.689) | -1.83 (7.852)
Statistical Analysis 1: Comparison: Levomilnacipran vs Quetiapine; Test type: Superiority; p = 0.913, t-test, 2 sided; Mean Difference (Final Values) = -0.236, 95% CI 2-sided [-4.559 to 4.088], Standard Error of Mean 2.158

11. Secondary Outcome: Changes in Sexual Dysfunction by Changes in Scores on Arizona Sexual Experience Scale (ASEX)
Description: ASEX is scale for sexual dysfunction to assess safety and tolerability of medication. Total scores range from 5-30. Higher scores indicate greater sexual dysfunction.
Time Frame: Baseline to Week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Levomilnacipran | Quetiapine
Number analyzed (Participants) | 29 | 30
score on a scale | -0.76 (2.923) | -0.30 (4.829)
Statistical Analysis 1: Comparison: Levomilnacipran vs Quetiapine; Test type: Superiority; p = 0.660, t-test, 2 sided; Mean Difference (Final Values) = -0.459, 95% CI 2-sided [-2.540 to 1.623], Standard Error of Mean 1.035

ADVERSE EVENTS:
Time Frame: Screening to Week 9
Arm/Group | Levomilnacipran | Quetiapine
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/31
Other Adverse Events (participants affected / at risk) | 16/29 | 22/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Levomilnacipran (N=29) | Quetiapine (N=31)
Nausea (Gastrointestinal disorders) | 4 | 4
Increase Appetite (General disorders) | 0 | 3
Weight Gain (General disorders) | 1 | 3
Weight Loss (General disorders) | 1 | 0
Headache (Nervous system disorders) | 6 | 2
Drowsiness (Nervous system disorders) | 2 | 12
Dizziness (Nervous system disorders) | 0 | 1
Confusion (Nervous system disorders) | 0 | 2
Dysuria (Renal and urinary disorders) | 2 | 0
Dry Mouth (General disorders) | 0 | 1
Sweating (General disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-18): https://cdn.clinicaltrials.gov/large-docs/98/NCT02720198/Prot_SAP_000.pdf